CLINICAL TRIAL: NCT02009228
Title: Single-Port Compared With Conventional Laparoscopic Cystectomy for Ovarian Dermoid Cysts
Brief Title: Single-port LC Might be Preferable for Managing Ovarian Dermoid Cyst.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, vghtpe user, Yi-Jen, Chen, M.D., Ph D., Department of Obstetrics and Gynecology, Taipei Veterans General Hospital, Taipei Veterans General Hospital, Taiwan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-06-004IA
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Abdominal Pain; Ovarian Spillage; Endobag Rupture; Ovarian Reserve
Keywords: Single-port laparoscopy; Abdominal pain; Ovarian spillage; Endobag rupture; Ovarian reserve
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-port laparoscopy (Active Comparator): The three-channel single-port: a 1.5-cm horizontal intraumbilical skin incision, a 1.5-cm to 2-cm rectus fasciotomy to open the peritoneal cavity, and the insertion of an Alexis small wound retractor (Applied Medical, Rancho Santa Margarita, CA). The wrist portion of a size 6.5 surgical glove was fixed to the outer ring of the wound retractor. A 12-mm trocar was inserted through a small hole made in one of the fingertips of the glove and advanced into the abdominal cavity. Two additional holes for the accessory channels were made in another fingertip of the glove, and two conventional 5-mm trocars were inserted through the holes.
  Interventions: Procedure: Ovarian cystectomy
- Conventional laparoscopy (Active Comparator): The 12-mm main troca was inserted via subumbilical incision after fully insufflation by verness needle and other 3 working 5-mm trocas were inserted under vision at right middle abdominal, left middle abdominal and suprapubic incisions.
  Interventions: Procedure: Ovarian cystectomy

INTERVENTIONS:
Procedure: Ovarian cystectomy
  Other Names: Dermoid cyst

SUMMARY:
Minimally invasive surgery has become the standard treatment for many gynecologic disease processes. In the last decade, numerous studies have demonstrated that laparoscopic approaches to various gynecologic oncology conditions-particularly for early-stage endometrial and cervical cancers as well as select pelvic masses-is feasible and results in shorter hospital stays, improved quality of life and comparable surgical and oncologic outcomes to abdominal staging.For instance, the typical gynecologic robotic surgical procedure will require Two to three 5-mm ports and one 12-mm laparoscopic ports. Recently, an even less invasive alternative to conventional laparoscopy surgery has been developed: laparoendoscopic single-site surgery (LESS), also known as single-port surgery. Single port laparoscopy is an attempt to further enhance the cosmetic benefits of minimally invasive surgery while minimizing the potential morbidity associated with multiple incisions. Preliminary advances in LESS as applied to urologic and gastrointestinal surgery demonstrate that the techniques are feasible provided that both optimal surgical technical expertise with advanced skills and optimal instrumentation are available. Recently, several publication showed the single port laparoscopic surgery is feasibility in gynecologic surgery including oophorectomy, cystecomty, and myomecomty. To our knowledge, the sample size of recent publication about single port surgery including cystectomy and myomecomty is small. Furthermore, these studies lack the comparison of single port and convectional laparoscopic surgery. Base on our recent study demonstrated that either the single-port or the conventional approach can be used for LAVH, but the single-port LAVH technique yielded less postoperative pain (Chen et al., Obestet Gynecol, 2011). The purpose of this study was to assess the feasibility of single port laparoscopic surgery in the treatment of benign gynecologic disease.

DETAILED DESCRIPTION:
This study was designed as a retrospective case-control study, and port placement was one of the differences in operative procedures between the two groups. Patients with ovarian dermoid cysts were evaluated at Taipei Veterans General Hospital from June 13, 2011 through June 12, 2013. Approval for the study was obtained from the hospital's ethics committee, and informed consent was obtained from all patients (VGHIRB 2011-06-004IA).

ELIGIBILITY:
Inclusion Criteria:

* the patient received cystectomy for ovarian dermoid cysts (even while pregnant), the cyst received an American Society of Anesthesiologists physical status classification of I or II, and the patient provided signed informed consent.

Exclusion Criteria:

* patients who received an oophorectomy for dermoid cyst or had a dermoid ovarian cyst with malignant potential and concomitant surgeries for uterine lesion, pelvic organ prolapse or urodynamic urinary incontinence were excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The outcome measures and ovarian reserve between single-port and conventional laparoscopic cystectomy in managing ovarian dermoid cysts. | The first 48 hours and 4 weeks after the surgery
  The outcome measures included operative time, blood loss, postoperative pain, and analgesic use in the first 48 hours after surgery.

SECONDARY OUTCOMES:
Ovarian reserve were compared with single-port and conventional laparoscopic cystectomy in managing ovarian dermoid cysts. | Before and 4 weeks after surgery.
  Ovarian reserve markers include serum estrogen (E2), follicle-stimulating hormone (FSH), luteinizing hormone (LH), and anti-Mullerian hormone (AMH) before and 4 weeks after surgery.

OTHER OUTCOMES:
Ovarian spillage and endobag rupture rates were compared between single-port and conventional laparoscopic cystectomy in managing ovarian dermoid cysts. | During operation.
  The ovarian spillage and endobag rupture rates were compared between single-port and conventional laparoscopic cystectomy in managing ovarian dermoid cysts during operation.

CONTACTS AND LOCATIONS:
Overall Officials: Ben-Shian Huang, M.D., Principal Investigator — Taipei Veterans General Hospital, National Yang Ming University Hosiptal, Ilan, Taiwan; Yi-Jen Chen, M.D., Ph D., Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veteran General Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Result] Chen YJ, Wang PH, Ocampo EJ, Twu NF, Yen MS, Chao KC. Single-port compared with conventional laparoscopic-assisted vaginal hysterectomy: a randomized controlled trial. Obstet Gynecol. 2011 Apr;117(4):906-912. doi: 10.1097/AOG.0b013e31820c666a. PMID 21422864